CLINICAL TRIAL: NCT05570357
Title: The Effects of Berberine and Cinnamon Supplementation on Diabetes Mangement
Brief Title: Berberine and Cinnamon in Management of Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Prof., National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 996401
Record Dates: First submitted 2022-10-02; First posted 2022-10-06 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Diabetes
Keywords: Diabetes; Berberine; Cinnamon
MeSH Terms: conditions — Diabetes Mellitus | interventions — tyramine-deoxysorbitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Dietary Supplement: Berberine+Cinnamon (TDS)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo (TDS)

INTERVENTIONS:
Dietary Supplement: Berberine+Cinnamon (TDS) — The supplements contains 400 mg Berberine, and 200 mg Cinnamon extract
  Arms: Intervention
Other: Placebo (TDS) — Placebo contains Maltodexterin
  Arms: Placebo

SUMMARY:
In this randomized clinical trial, patients with diabetes will be randomly assigned to receive either Berberine, and Cinnamon supplements or placebo for 12 weeks. Then the glycemic characteristics will be compared in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-70 years
* Diagnosed type-2 diabetes mellitus (based on American Diabetes Association criteria)

Exclusion Criteria:

* Patients with an allergy to berberine /cinamon

  * Lactation, pregnancy
  * Patients with any malignancy
  * Patients with unrelated chronic illness
  * Patients with cardiac, liver or respiratory failure

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
HbA1C | 0 and 12th week
  HbA1C change from baseline

SECONDARY OUTCOMES:
Fasting blood sugar | 0 and 12th week
  Blood sugar change from baseline
Lipid profile | 0 and 12th week
  lipid profiles change from baseline
Anthropometric measurements | 0 and 12th week
  weight, height, BMI, WC
Blood Pressure | 0 and 12th week
  measuring according to the BP measurement guideline
CRP | 0 and 12th week
  measuring the blood concentration of C-reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- Azita Hekmatdoost, Tehran, Middle East, Iran

IPD SHARING:
Plan to Share IPD: Undecided